CLINICAL TRIAL: NCT03950492
Title: Feasibility of Deep Brain Stimulation as a Novel Treatment for Refractory
Brief Title: Feasibility of Deep Brain Stimulation as a Novel Treatment for Refractory Opioid Use Disorder
Acronym: DBS_OUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Medtronic (Industry)
Responsible Party: Principal Investigator, Ali Rezai, Principal Investigator, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1903499841; 1UG3DA047714-01 (NIH)
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Opioid-Related Disorders
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is an open-label, safety, tolerability, and feasibility study for participants who have treatment refractory OUD that are eligible to have deep brain stimulation (DBS) targeting the NAc/VC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- OUD DBS (Experimental): This is a single arm study. Participants will be followed in an inpatient service for two weeks to gather baseline data followed by DBS placement and up to 6 weeks inpatient for clinical stabilization and DBS titration. All participants will then be followed twice a week for 12 weeks in the outpatient setting and then once a week for a total of 52 weeks post-titration.
  Interventions: Device: Deep Brain Simulator

INTERVENTIONS:
Device: Deep Brain Simulator — This is an open-label, safety, tolerability, and feasibility study for participants who have treatment refractory OUD that are eligible to have DBS targeting the NAc/VC.

SUMMARY:
The purpose of this clinical study is to investigate the safety, tolerability, and feasibility of Deep Brain Stimulation (DBS) of the nucleus accumbens (NAc) and ventral internal capsule (VC) for participants with treatment refractory opioid use disorder (OUD) who have cognitive, behavioral, and functional disability. This study will also provide critical information for planning subsequent clinical trials.

DETAILED DESCRIPTION:
The overarching goal of this study is to evaluate the safety, tolerability, feasibility and impact on outcomes of NAc/VC DBS for treatment refractory OUD. In treatment refractory OUD, innovative approaches and more invasive interventions including DBS are warranted to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills current DSM-5 (American Psychiatric Association Diagnostic and statistical manual of mental disorders, 5th ed, 2013) diagnostic criteria for OUD (severe) and at least a 5-year history.
* Participants may have comorbid SUD diagnoses at mild, moderate or severe levels, however OUD must be the primary disorder for which the individual is seeking treatment and the other use disorders must occur in the context of relapse
* Failed at least two levels of treatment (outpatient/Comprehensive Opioid Addiction Treatment (COAT), intensive outpatient/intensive COAT, residential, inpatient, Adult Intensive Outpatient Program (AIOP), Dual Diagnosis Unit (DDU), which included buprenorphine/naloxone.
* At least two overdose survivals or one overdose survival and one life-threatening infectious disease complication with relapse after treatment (e.g., endocarditis with valve repair/replacement) within the past 1 year.
* Family/Social Support/Involvement (as assessed via the Multidimensional Scale of Perceived Social Support).
* Is able to provide informed consent.

Exclusion Criteria:

* Medical problems requiring intensive medical or diagnostic management.
* Diagnosis of acute myocardial infarction or cardiac arrest within the previous 6 months.
* History of a neurosurgical ablation procedure.
* Any medical contraindications to undergoing DBS surgery.
* History of hemorrhagic stroke.
* Life expectancy of <3 years
* Past or present diagnosis of schizophrenia, psychotic disorder, bipolar disorder, or untreated depression other than one determined to be substance induced (assessed via SCID-5). Any treated depression has to have been in remission for one year.
* Baseline assessment on the Hamilton Depression Rating Scale (HAMD) of greater than 17 or increased risk of suicide based upon any positive response on the Columbia Suicide Severity Scale.
* Cluster A or B Personality Disorders.
* Diagnosis of dementia.
* History of neurological disorder.
* History of previous neurosurgery (brain) or head trauma.
* History of suicide attempt.
* Parental history of completed suicide.
* Abnormal coagulation lab studies or uncontrolled hypertension.
* Implanted neurostimulators.
* Any current CNS infection or infection with the Human Immunodeficiency Virus (HIV).
* Unable to undergo MR-imaging.
* Documentation of MRI abnormality indicative of a neurological condition.
* Substance abuse treatment mandated by court of law.
* Pregnant or planning to become pregnant.
* Conditions requiring diathermy.
* Anticoagulant treatment.
* Primary language other than English.
* Any evidence of systemic infection.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Rezai, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezai AR, Mahoney JJ, Ranjan M, Haut MW, Zheng W, Lander LR, Berry JH, Farmer DL, Marton JL, Tirumalai P, Mears A, Thompson-Lake DGY, Finomore VS, D'Haese PF, Aklin WM, George DT, Corrigan JD, Hodder SL. Safety and feasibility clinical trial of nucleus accumbens deep brain stimulation for treatment-refractory opioid use disorder. J Neurosurg. 2023 Jun 9;140(1):231-239. doi: 10.3171/2023.4.JNS23114. Print 2024 Jan 1. PMID 37329519

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OUD DBS
Started | 4
Completed | 2
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | OUD DBS
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Study-Emergent Adverse Events
Description: Study participants will be closely monitored for adverse events following DBS surgery with regular check-ups by study personnel.
Time Frame: Enrollment - 52 weeks
Measure: Number; unit: Adverse Events
Arm/Group | OUD DBS
Number analyzed (Participants) | 4
Adverse Events
  Total Mild AEs | 74
  Mild AE - Unexpected | 32
  Mild AE- Expected | 42
  Total Moderate AEs | 29
  Moderate AE - Unexpected | 20
  Moderate AE - Expected | 9
  Total Severe AEs | 5
  Severe AE - Unexpected | 4
  Severe AE - Expected | 1
  Mild AE - Definitely Related (Surgical Procedure) | 1
  Mild AE - Definitely Related (Disorder) | 1
  Mild AE - Probably Related (Surgical Procedure/Stimulation) | 1
  Mild AE - Probably Related (Stimulation) | 2
  Mild AE - Probably Related (Disorder) | 30
  Mild AE - Possibly Related (Stimulation/Disorder) | 4
  Mild AE - Possibly Related (Stimulation) | 1
  Mild AE - Possibly Related (Disorder) | 1
  Mild AE - Unlikely Related | 6
  Mild AE - Unrelated | 27
  Moderate AE - Probably Related (Surgical Procedure) | 1
  Moderate AE - Probably Related (Stimulation/Disorder) | 1
  Moderate AE - Probably Related (Disorder) | 5
  Moderate AE - Possibly Related (Disorder) | 1
  Moderate AE - Unlikely Related | 1
  Moderate AE - Unrelated | 20
  Severe AE - Unlikely Related | 2
  Severe AE - Possibly Related (Surgical Procedure) | 1
  Severe AE - Possibly Related (Disorder) | 2

2. Primary Outcome: Change in Opioid Use
Description: Opioid use as measured by quantitative urine toxicology via high pressure liquid chromatography.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | OUD DBS
Number analyzed (Participants) | 4
participants
  Number of Participant's Opioid Negative through 12 Week Endpoint | 2
  Number of Participant's Opioid Positive through 12 Week Endpoint | 2

3. Secondary Outcome: Participant Survival
Description: Incidence of drug overdose deaths among the participants.
Time Frame: 12 -52 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Treatment Retention
Description: Participants' retention in traditional medication assisted treatment (MAT).
Time Frame: 12 - 52 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Serious Infectious Disease Complications
Description: Laboratory tests and evaluation to discern presentation of infectious disease.
Time Frame: 12 - 52 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Mood, Craving and Executive Function
Description: Participants will complete standardized measures of mood, drug craving, and executive function at 12 weeks and 24 weeks post DBS titration.
Time Frame: 12 and 24 weeks post surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Frontal Lobe Metabolism
Description: 18fluoro-Deoxy-Glucose (FDG) PET will be use to determine if there is an increase in frontal lobe metabolism following DBS
Time Frame: 3 weeks and 12 weeks post surgery
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Dopamine
Description: C11 Raclopride PET may be used to examine for changes in dopamine at 12 weeks post titration.
Time Frame: 3 weeks and 12 weeks post surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Participants were evaluated for AEs from the time consent was obtained until study closure or study exit. AEs were assessed at each visit and via self-report. The following were not considered AEs:
  Inefficient DBS reprogramming Temporary stimulation-related effects during programming Expected postoperative symptoms, unless significant Worsened pre-existing conditions Unrelated medical/surgical procedures Routine battery replacement Non-medically significant technical observations/events
Groups:
- OUD DBS: This is a single arm study. Participants will be followed in an inpatient service for two weeks to gather baseline data followed by DBS placement and up to 6 weeks inpatient for clinical stabilization and DBS titration. All participants will then be followed twice a week for 12 weeks in the outpatient setting and then once a week for a total of 52 weeks post-titration.
  Deep Brain Stimulator: This is an open-label, safety, tolerability, and feasibility study for participants who have treatment refractory OUD that are eligible to have DBS targeting the NAc/VC.
Arm/Group | OUD DBS
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OUD DBS (N=4)
Relapse of Opioid Use (Psychiatric disorders) | 1 (1)
Blacked Out (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OUD DBS (N=4)
Abnormal TEG (Blood and lymphatic system disorders) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 1 (2)
Hypotension (Cardiac disorders) | 1 (4)
Palpitations (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
GI Disorders, Other - Decreased Appetite (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (5)
Sick feeling (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Acute pharyngitis (sore throat) (General disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Dysgeusia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (10)
Headache (General disorders) | 2 (7)
Insomnia (General disorders) | 3 (5)
Lethargy (General disorders) | 1 (3)
Malaise (General disorders) | 1 (1)
Motor vehicle accident (General disorders) | 1 (1)
Nasal Congestion (General disorders) | 1 (2)
Pharyngitis (General disorders) | 1 (1)
Restlessness (General disorders) | 1 (5)
Sweats (General disorders) | 1 (3)
Tremor (General disorders) | 1 (2)
Twitching left eye brow (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Dental pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mouth pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain- Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Sprain, left ankle (Musculoskeletal and connective tissue disorders) | 1 (1)
Tooth Ache (Musculoskeletal and connective tissue disorders) | 1 (2)
Toothache (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic Migraine (Nervous system disorders) | 1 (1)
Fatigue (Nervous system disorders) | 1 (1)
Hypoxia (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Auditory Hallucinations (Psychiatric disorders) | 1 (1)
Blacked out (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Overuse-no adverse effect-Suboxone misuse (Psychiatric disorders) | 1 (1)
Relapse (Psychiatric disorders) | 1 (1)
Sleep Disturbance (Nightmares) (Psychiatric disorders) | 1 (1)
Sleep Disturbances, Nightmares (Psychiatric disorders) | 1 (1)
Bacteria Urine (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Renal Calculi (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abrasion, right wrist (Skin and subcutaneous tissue disorders) | 1 (1)
Bilateral Foot Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising (arm) (Skin and subcutaneous tissue disorders) | 1 (1)
Burn (Skin and subcutaneous tissue disorders) | 1 (1)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Infusion Site Irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Injury, Other - Physical Altercation with bruising, edema, pain (Skin and subcutaneous tissue disorders) | 1 (1)
Laceration (chin) (Skin and subcutaneous tissue disorders) | 1 (1)
Papular urticaria - bug bites left ankle (Skin and subcutaneous tissue disorders) | 1 (1)
Parasthesia, left ear (Skin and subcutaneous tissue disorders) | 1 (1)
Paresthesia - Hand (Skin and subcutaneous tissue disorders) | 1 (1)
Penile rash (Skin and subcutaneous tissue disorders) | 1 (1)
Poison Ivy (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Macro-Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, facial (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Wound - insect bite right leg (Skin and subcutaneous tissue disorders) | 1 (1)
Incarceration (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT03950492/Prot_SAP_000.pdf